CLINICAL TRIAL: NCT01744431
Title: Can Thrombin Generation Measurement Predict the Risk of Venous Thromboembolism in Acute Ill Patients
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Elias mazen, Director of Internal Medicine, HaEmek Medical Center, Israel
Other Study IDs: thrombin generation
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
Can thrombin generation measurement predict the risk of venous thromboembolism in acute ill patients

Traditional coagulation tests do not assess the whole coagulation system. Thrombin generation assays measure the ability of plasma sample to generate thrombin following in vitro activation of coagulation. In contrast to the classical clotting assays, thrombin generation reflects and integrates all pro and anticoagulant reactions that regulate the formation and inhibition of thrombin.

The aim of our study is to investigate whether thrombin generation would be able to predict a hypercoagulable state in acute ill patients admitted in the internal medical departments and how it correlates with the Padua prediction score, a score that could assists the risk for venous thromboembolism in hospitalized medical patients.

In total 300 patients are planned for inclusion in this trial. After signing an informed consent a blood sample will be obtained from each participant. We will measure the thrombin generation over time in plasma assessed by the calibrated automated thrombogram (CAT).

ELIGIBILITY:
Inclusion Criteria:

* signed inform consent

Exclusion Criteria:

* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
venous thromboembolism | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: mazen elias, MD, Principal Investigator — Emek Medical Center
Locations (1):
- Emek medical center, Afula, Israel